CLINICAL TRIAL: NCT00685230
Title: Prospective, Randomized, Double-Blind, Controlled Study of Alacramyn® vs. Placebo in Pediatric Patients With Systemic Signs of Scorpion Sting Envenomation
Brief Title: Double-Blind, Alacramyn® vs. Placebo in Pediatric Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Collaborators: University of Arizona (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Dr. Walter Garcia Ubbelohde/Clinical Research Manager, Instituto Bioclon
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL-02/03
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Scorpion Sting Envenomation
Keywords: scorpion sting; envenomation; alacramyn
MeSH Terms: conditions — Scorpion Stings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Alacramyn and midazolam as needed
  Interventions: Biological: Antivenin Centruroides (scorpion) equine immune F(ab)2
- 2 (Placebo Comparator): placebo and midazolam as needed
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Antivenin Centruroides (scorpion) equine immune F(ab)2 — 3 vials of Alacramyn reconstitued in 50 ml of normal saline as a IV infusion over 10 minutes.
  Other Names: Anascorp
  Arms: 1
Other: Placebo — Placebo reconstituted in 50 ml of normal saline administered over 10 min
  Arms: 2

SUMMARY:
There is no FDA approved therapy for the treatment of scorpion envenomation, Centruroides scorpion envenomation produces a pattern of neurotoxicity with a spectrum of severity ranging from trivial to life threatening. Patients stung by Centruroides scorpions develop a clinical syndrome which may require sedation with benzodiazepines and observation for 6 to 28 hours of intensive care monitoring. A safe therapy is necessary to halt the progression of symptoms early in the clinical course while avoiding the clinical deterioration that can occur en route to a tertiary facility. Alacramyn® is anticipated to be safer and more effective than the present standard of care, midazolam, and faster-acting such that the need for transport of most rural patients will be eliminated and will reduce hospitalization time.

The working hypotheses are as follows:

1. The investigational antivenom is safe as treatment of scorpion sting envenomation.
2. The investigational antivenom is effective as treatment of scorpion sting envenomation.

DETAILED DESCRIPTION:
The purpose of this Prospective, Randomized, Double-Blind, Controlled, Multicenter Treatment Protocol, phase III trial is to examine the safety and efficacy of Alacramyn® for treatment of patients envenomed by scorpion sting.

This study will take place in two pediatric Intensive care units in Tucson, Arizona.

Patients who arrive at the emergency clinic presenting with scorpion sting symptoms will be evaluated for treatment with respect to the inclusion/exclusion criteria according to the study procedures. Only patients with clinically important systemic signs of scorpion sting envenomation will be included in the study. Baseline measures will include severity evaluation of the scorpion sting envenomation. The patient's vital signs, concomitant medication, medical history and demographic data will be collected. Blood tests will be done for haematology, chemistry, venom and anti-venom levels and urine test.

After informed consent and inclusion7exclusion criteria have been obtained and verified, and the baseline measurements have been done, three vials of Alacramyn® or placebo will be administered. During the following 3 hours, midazolam will continue, if indicated for control of agitation.

Patients off midazolam sedation after receiving study drug and no longer manifesting clinically important systemic signs of scorpion envenomation will be discharge at 4 hours, or 2 hours following cessation of midazolam drip, whichever occurs later. Prior to discharge repeat lab work, physical assessments, and vital signs will be done. Patients still requiring midazolam sedation and/or manifesting clinically important systemic signs of scorpion envenomation will be treated with standard of care for the duration of clinical symptoms. Those remaining for extended care undergo final study assessments at time of hospital discharge or at 24 hours after study drug infusion if hospitalization continues.

All patients who participated in the study will be contacted 7 and 14 days after treatment, looking for symptoms suggestive of ongoing venom effect, delayed serum sickness as well as for any other adverse event reported by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of 6 months to 18 years of age
* Presenting for emergency treatment within 5 hours with clinically important systemic signs of scorpion sting envenomation.
* Signed written Informed Consent by patient or legal guardian.
* No participation in a clinical drug trial within the last month or concomitantly.

Exclusion Criteria:

* Allergy to horse serum.
* Use within the past 24 hours of drugs expected to alter immune response: H1 or H2 blockers, corticosteroids.
* Use of any antivenom within the last month or concomitantly.
* Underlying medical conditions that significantly alter immune response: bone marrow suppression congenital or acquired immuno-deficiency state, chemotherapy and chronic corticosteroid use.
* Allergy to midazolam.
* More than 0.3mg/kg of body weight of midazolam administered during the hour prior to study drug infusion.
* Concurrent medical condition involving a baseline neurologic status mimicking envenomation (chorea, tardive dyskinesia, uncontrolled epilepsy).
* Pregnant and nursing women.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2004-05; Primary Completion 2005-08 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary study endpoint is the resolution of clinically important signs of scorpion envenomation | 4 hours

SECONDARY OUTCOMES:
Alacramyn®-treated patients require significantly less benzodiazepine sedation than placebo controls, for control of agitation | 4 hours
Venom blood levels decrease after Alacramyn® treatment, while the placebo group continues to have elevated blood venom levels | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Boyer, MD, Principal Investigator — Poison and Drug Center; Walter Garcia, MD, Study Director — Instituto Bioclon S.A. de C.V.; Alejandro Alagon, PhD, Study Chair — Universidad Nacional Autonoma de Mexico
Locations (2):
- United States (2):
  - Tucson Medical Center, Tucson, Arizona
  - University Medical Center, Tucson, Arizona

REFERENCES:
- [Background] Likes K, Banner W Jr, Chavez M. Centruroides exilicauda envenomation in Arizona. West J Med. 1984 Nov;141(5):634-7. PMID 6516334
- [Background] Connor, D.A., Seldon, B.S., Scorpion Envenomation. Chapter in Wilderness Medicine; Management of Wilderness and Environmental Emergencies. 3rd edition. Auerbach PS, ed., Mosby Yearbook, Inc. St. Louis, MO. pp 831-842
- [Background] Gibly R, Williams M, Walter FG, McNally J, Conroy C, Berg RA. Continuous intravenous midazolam infusion for Centruroides exilicauda scorpion envenomation. Ann Emerg Med. 1999 Nov;34(5):620-5. doi: 10.1016/s0196-0644(99)70164-2. PMID 10533010
- [Background] Curry SC, Vance MV, Ryan PJ, Kunkel DB, Northey WT. Envenomation by the scorpion Centruroides sculpturatus. J Toxicol Clin Toxicol. 1983-1984;21(4-5):417-49. doi: 10.3109/15563658308990433. PMID 6381751
- [Background] Chavez-Haro A., Gonzalez J., Paniagua nJ., Efficiency and Security Comparison between Two Different Scorpion-derived Antivenom in Mexico, Abstract, Leon Study Data Analysis.
- [Background] Gonzalez, C., et al, Development of an Immunoenzymatic Assay for the Quantification of Scorpion Venom in Plasma, Abstract, Cuernavaca, 2000
- [Background] LoVecchio F, Welch S, Klemens J, Curry SC, Thomas R. Incidence of immediate and delayed hypersensitivity to Centruroides antivenom. Ann Emerg Med. 1999 Nov;34(5):615-9. doi: 10.1016/s0196-0644(99)70176-9. PMID 10533009
- [Background] Alagon Cano, A., Gozalez Juarez, C., From Serotherapy to Fabotherapy, Abstract, Cuernavaca, 1998.
- [Background] Cabral-Soto, J., et al, Comparison of Efficacy between Two Antiscorpion Antivenoms, Abstract, Cuernavaca, 2000, Clinical Study Report, Randomized, Double-Blind, Variable dosing of Alacramyn in Patients With Scorpion Sting (this was done with two approved products in Mexico, Alacramyn and Birmex), March 2002.
- [Background] Madrazo Navarro, M., et al, Animales Ponzoñosos en la Población Derechohabiente del IMSS 1990-1996.
- [Background] Dart, R.C., Horowitz, R.S., Use of Antibodies as Antivenoms: A primitive Solution for Complex Problem? Rocky Mountain Poison and Drug Center, Denver Co, USA.
- [Background] TESS Data Collection Manual (available upon request)
- [Background] Berg RA, Tarantino MD. Envenomation by the scorpion Centruroides exilicauda (C sculpturatus): severe and unusual manifestations. Pediatrics. 1991 Jun;87(6):930-3. No abstract available. PMID 2034501
- [Background] Rachesky IJ, Banner W Jr, Dansky J, Tong T. Treatments for Centruroides exilicauda envenomation. Am J Dis Child. 1984 Dec;138(12):1136-9. doi: 10.1001/archpedi.1984.02140500042015. PMID 6507396
- [Background] Rimsza ME, Zimmerman DR, Bergeson PS. Scorpion envenomation. Pediatrics. 1980 Aug;66(2):298-302. PMID 7402816
- [Derived] Boyer LV, Theodorou AA, Berg RA, Mallie J; Arizona Envenomation Investigators; Chavez-Mendez A, Garcia-Ubbelohde W, Hardiman S, Alagon A. Antivenom for critically ill children with neurotoxicity from scorpion stings. N Engl J Med. 2009 May 14;360(20):2090-8. doi: 10.1056/NEJMoa0808455. PMID 19439743
- See also: The University of Arizona — http://www.arizona.edu/
- See also: Instituto de Biotecnologia de la UNAM — http://www.ibt.unam.mx